CLINICAL TRIAL: NCT00979732
Title: Randomized, Double-blind, Placebo-controlled Trial to Investigate the Effect of Grape Seed Extract Delivered in a Beverage on Blood Pressure in Individuals With Pre-hypertension.
Brief Title: The Effect of Grape Seed Extract on Blood Pressure in People With Pre-Hypertension
Acronym: GSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Polyphenolics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSE 2009-050
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: high blood pressure; dietary supplements; nutrition
MeSH Terms: conditions — Hypertension | interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSE beverage active (Active Comparator): grape seed extract beverage 150 mg/BID
  Interventions: Dietary Supplement: grape seed extract
- GSE beverage placebo (Placebo Comparator): grape seed extract placebo beverage 150 mg/BID
  Interventions: Dietary Supplement: grape seed extract placebo

INTERVENTIONS:
Dietary Supplement: grape seed extract — grape seed extract 150 mg twice a day (BID) in beverage or capsule form
  Arms: GSE beverage active
Dietary Supplement: grape seed extract placebo — grape seed extract 150 mg twice a day (BID) in beverage or capsule form
  Arms: GSE beverage placebo

SUMMARY:
In this research study, the investigators are interested in learning how extracts from grape seeds can help those individuals with high blood pressure. The investigators also hope to learn how grape seed extract effects your blood and cell functions.

The grape seed extract the investigators will use in the study will be provided either in a beverage or a capsule form and is currently available on the market. This study is also using a placebo; therefore the treatment subjects receive may or may not contain the grape seed extract.

The purpose of this study is to determine if the grape seed extract (GSE) will lower blood pressure in people with slightly high blood pressure (Pre-Hypertension).

DETAILED DESCRIPTION:
Elevated blood pressure, or hypertension, is a major risk factor for heart disease and stroke. Systolic and diastolic blood pressures meeting criteria for "pre-hypertension" double the absolute risk of stroke and ischemic heart disease over an extended age range from the 4th to the 8th decade of life. Lifestyle, particularly the diet, is critical in the prevention and management of hypertension. Polyphenolic compounds from various plant foods can promote blood pressure regulation and vascular health through protection of the endothelium from oxidant and or inflammatory stress and or stimulation of smooth muscle relaxation.

We will use a purified grape seed extract (GSE) in the proposed trial. This extract has been granted Generally Recognized as Safe (GRAS) status by Food and drug administration (GRAS Notice # GRN 000125, dated 08/18/2003, FDA, USA). Furthermore, GSE for use in the present trial has been used in previous human clinical trails and shown potent vasodilator properties in vitro and blood pressure lowering in metabolic syndrome patients. The proposed trial aims to verify the blood pressure lowering effect of GSE in an 'at risk' population for hypertension and to explore the extent to which other pathways of chronic disease may be modulated by GSE consumption.

Given this, the objectives of this study are as follows:

1. The primary objective of the proposed study is to demonstrate the effectiveness of GSE to lower blood pressure in pre-hypertensive individuals.
2. Secondary objectives will investigate the role of GSE to improve inflammatory- and oxidative stress- status, as well as its effect on endothelium function.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* pre-hypertensive

  * systolic blood pressure (mmHg) 120 - 139 or
  * diastolic blood pressure (mmHg) 80 -89
* no clinical evidence of cardiovascular, respiratory, renal, gastrointestinal or hepatic disease

Exclusion Criteria:

* pregnant and or lactating
* taking over the counter antioxidant supplements
* taking prescription medications that may interfere with study procedures or endpoints
* unusual dietary habits
* actively trying to lose or gain weight
* addicted to drugs and/or alcohol
* medically documented psychiatric or neurological disturbances
* smoker (past smoker may be allowed if cessation is > 2 years)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11-15 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2014-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, PhD, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology; Indika Edirisinghe, PhD, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edirisinghe I, Burton-Freeman B, Tissa Kappagoda C. Mechanism of the endothelium-dependent relaxation evoked by a grape seed extract. Clin Sci (Lond). 2008 Feb;114(4):331-7. doi: 10.1042/CS20070264. PMID 17927567
- [Background] Brahmesh S, Edirisinghe I, Randolph J, Steinberg F and Kappagoda T. Effect of a polyphenoics extracts of grape seeds (GSE) on blood pressure in patients with metabolic syndrome (MetS). FASEBJ. 2006;20:A305.
- [Background] Sivaprakasapillai B, Edirisinghe I, Randolph J, Steinberg F, Kappagoda T. Effect of grape seed extract on blood pressure in subjects with the metabolic syndrome. Metabolism. 2009 Dec;58(12):1743-6. doi: 10.1016/j.metabol.2009.05.030. Epub 2009 Jul 15. PMID 19608210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at the Clinical Nutrition Research Center at the Illinois Institute of Technology (Chicago, IL, USA) from 2010 to 2014.
Pre-assignment Details: Eligible subjects started with a 2-week run-in period drinking the Placebo beverage twice per day. After the 2-week run-in period, subjects were randomised to one of the two groups (Placebo or GSE beverage), equally allocated to each treatment (1:1 randomisation ratio).
Period: Overall Study
Arm/Group | GSE Beverage Active | GSE Beverage Placebo
Started | 15 | 18
Completed | 12 | 17
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were collected at the screening
Groups:
- Total: Total of all reporting groups
Arm/Group | GSE Beverage Active | GSE Beverage Placebo | Total
Number analyzed (Participants) | 12 | 17 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10) | 42 (10) | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 11 | 15 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: BP was monitored using ambulatory BP monitors (Ambulo2400; Tiba Medical, Inc.) that were programmed to take BP measurements automatically at 1-h intervals for a period of 24 h. BP measurements were scheduled at week 0 and 6 of the intervention (for efficacy assessment). Day-time BP and night-time BP were divided based on the subject's sleeping hours and hours awake.
Time Frame: 6 weeks
Population: All completers
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | GSE Beverage Active | GSE Beverage Placebo
Number analyzed (Participants) | 12 | 17
mmHg | 118 (2.3) | 127 (1.9)

2. Secondary Outcome: Plasma Insulin Level Over 6 Weeks
Description: After 10-12 h of overnight fasting, fasting blood samples were collected at week 0 (baseline) and week 3 and 6 of the intervention. plasma insulin were evaluated.
Time Frame: 6 weeks
Population: All completer
Measure: Mean (Standard Error); unit: µIU/mL
Arm/Group | GSE Beverage Active | GSE Beverage Placebo
Number analyzed (Participants) | 12 | 17
µIU/mL | 17.8 (1.5) | 20.9 (1.2)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | GSE Beverage Active | GSE Beverage Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 0/12 | 0/17

LIMITATIONS AND CAVEATS:
The study was not sufficiently powered to detect significant differences on the secondary end points. We observed large inter-individual variability in plasma phenolic concentrations, requiring a greater sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No